CLINICAL TRIAL: NCT05818462
Title: Effect of Pelvic Radiation Therapy on the Urinary and Musculoskeletal Systems of Survivors of Childhood Cancer
Brief Title: Bladder and Bone Effects of Pelvic Radiation Therapy in Childhood Cancer Survivors
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 22-1533.cc
Record Dates: First submitted 2023-03-09; First posted 2023-04-18 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Childhood Cancer
MeSH Terms: conditions — Neoplasms | interventions — Urinalysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who received EBRT to the pelvis.: Childhood cancer survivors who were treated with chemotherapy and radiation therapy to the pelvis, with or without surgical intervention. This group will consist of both primary pelvic sarcomas as well as patients who received whole abdominal radiation that included bladder exposure.
  Interventions: Diagnostic Test: Uroflow testing; Diagnostic Test: Bladder Scan; Other: Dysfunctional Voiding Scoring System Survey; Diagnostic Test: DEXA Scan of pelvis and sacral spine; Diagnostic Test: Urine tests for specific biomarkers
- Control cohort.: Childhood cancer survivors who have been treated for a sarcoma who did not receive pelvic radiation, and were treated with chemotherapy, with or without surgical intervention or radiation therapy (outside of the pelvis). These patients will be matched as closely as possible to Group 1 to match chemotherapy regimens, and sex.
  Interventions: Diagnostic Test: Uroflow testing; Diagnostic Test: Bladder Scan; Other: Dysfunctional Voiding Scoring System Survey; Diagnostic Test: DEXA Scan of pelvis and sacral spine; Diagnostic Test: Urine tests for specific biomarkers

INTERVENTIONS:
Diagnostic Test: Uroflow testing — Uroflowmetry is a test that measures the volume of urine released from the body, the speed with which it is released, and how long the release takes.
Diagnostic Test: Bladder Scan — Bladder scan measures ultrasonic reflections within the patient's body to differentiate the urinary bladder from the surrounding tissue. In this case, it is used to detect the volume of urine in the bladder.
Other: Dysfunctional Voiding Scoring System Survey — The Dysfunctional Voiding Symptom Score to provide accurate and objective numerical, grading of voiding behaviors of children.
Diagnostic Test: DEXA Scan of pelvis and sacral spine — DEXA (dual x-ray absorptiometry) scans measure bone density (thickness and strength of bones) by passing a high and low energy x-ray beam (a form of ionizing radiation) through the body, usually in the hip and the spine.
Diagnostic Test: Urine tests for specific biomarkers — Urine tests for specific biomarkers (ATP, NGF, BNDF and urine proteomic screening).

SUMMARY:
The aim of this study is to measure and evaluate the effects of pelvic external beam radiation therapy (EBRT) on lower urinary tract (LUT) function and bone mineralization.

DETAILED DESCRIPTION:
The aim of this study is to measure and evaluate the effects of pelvic external beam radiation therapy (EBRT) on lower urinary tract (LUT) function and bone mineralization. The overarching hypothesis is that patients who received EBRT to the pelvis will have an increased rate of LUT dysfunction and osteoporosis even when controlled for chemotherapeutic exposures, using patients with similar chemotherapy regimens as controls. Between these two groups, the team expect to observe significant differences in both patient-reported outcomes and direct measures of LUT function.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age who were treated were diagnosed in 2007 or later and received chemotherapy for solid tumor malignancy, with completion of therapy (whether chemotherapy or radiation) at least one year prior to study enrollment.

Exclusion Criteria:

* Patients with known dysfunctional voiding prior to cancer treatment.
* Patients with tumor resection of bladder, prostate or gynecologic organs will be excluded.

Ages: 2 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cohort 1: Childhood cancer survivors who were treated with chemotherapy and radiation therapy to the pelvis, with or without surgical intervention. This group will consist of both primary pelvic sarcomas as well as patients who received whole abdominal radiation that included bladder exposure.
  Cohort 2: Childhood cancer survivors who have been treated for a sarcoma who did not receive pelvic radiation, and were treated with chemotherapy, with or without surgical intervention or radiation therapy (outside of the pelvis). These patients will be matched as closely as possible to Group 1 to match chemotherapy regimens, and sex.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Uroflow and Bladder Scan Results | 1.5 years
  aggregate measured by voiding time (seconds, s), total voided volume (mL), average uroflow rate (mL/s), maximum uroflow rate (mL/s), uroflow pattern or curve (bell-shaped, tower-shaped, staccato, interrupted or plateau), and post void residual (mL)

SECONDARY OUTCOMES:
DVSS Scores | 1.5 years
  2. Total DVSS survey scores to determine patient-reported urinary symptom. Gender-specific DVSS total score thresholds: males ≥9, females ≥6. Minimum DVSS score is 0 points. Maximum DVSS score is 30 points.
Number of Patients with Osteoporosis | 1.5 years
  4. Rates of osteopenia and osteoporosis, as determined by bone density Z-score using DEXA scan of pelvis and sacral spine. Osteopenia is defined as a z-score between - 1 to -2.5, while osteoporosis is defined as a z-score below -2.5
DEXA Scan Results | 1.5 years
  3. Average pelvic and sacral spine bone mineral density Z-scores, as determined by a DEXA scan of pelvis and sacral spine.

OTHER OUTCOMES:
Biomarker - ATP | 1.5 years
  Measure biomarker ATP in order to determine urinary biomarkers for investigation into radiation-induced LUTD.
Biomarker - NGF | 1.5 years
  Measure biomarker NGF in order to determine urinary biomarkers for investigation into radiation-induced LUTD.
Biomarker - BNDF | 1.5 years
  Measure biomarker BNDF in order to determine urinary biomarkers for investigation into radiation-induced LUTD.
Biomarker - urine proteomic screening results | 1.5 years
  Measure urinary excreted proteins and peptides via urine proteomic screening in order to determine urinary biomarkers for investigation into radiation-induced LUTD.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Edwards, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Colorado Research Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No